CLINICAL TRIAL: NCT00705497
Title: Radiofrequency Ablation of Tumors (RFA) A Phase I Study
Brief Title: Radiofrequency Ablation of Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RFA
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2011-06

CONDITIONS: Primary Tumors; Metastatic Tumors
Keywords: Radiofrequency tumor ablation; RFA
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Radiofrequency Tumor Ablation

INTERVENTIONS:
Procedure: Radiofrequency Tumor Ablation — Radiofrequency tumor ablation (RFA) is an imaging guided percutaneous or intra-operative procedure that uses a probe on the end of a sharp needle that is inserted directly into the tumor. The tumor is ablated by heating the probe (using electrical current alternating at radio frequency) which raises the temperature of the tumor potentially causing irreversible cell death.

SUMMARY:
Background: This prospective study was designed to be the first to evaluate the toxicity of radiofrequency ablation (RFA) in patients with recurrent pediatric solid tumors.

Methods: From 2003 through 2006, we conducted a phase I, IRB-approved study of RFA for recurrent solid tumors. A multidisciplinary cancer management team selected appropriate candidates for the study. Imaging-guided RFA was performed percutaneously. Response was assessed at 3 months. Repeat RFA was performed for some incompletely ablated or new lesions.

ELIGIBILITY:
Inclusion Criteria:

General

* Any age
* Previously diagnosed malignancy (including aggressive fibromatosis) originally acquired during childhood (<21 years-of-age)
* Patients who have undergone previous RFA may be enrolled again (different disease site) or receive subsequent ablation (same disease site) as long as the eligibility criteria are met at the time of re-enrollment, or a second ablation on study.
* The subject is medically appropriate for the study as determined by a consensus of professionals at multidisciplinary tumor conference prior to enrollment. This discussion will be documented in the chart of the potential subject to be recruited for this study.
* Histopathological material is available prior to the RF ablation except in patients with obvious tumor recurrence.
* No Pacemakers or Automatic Implantable Cardioverter/Defibrillators (AICDs)
* No tissue burns anticipated from implanted metal
* Normal renal function (Creatinine < 2mg/dL)
* Absolute neutrophil count (ANC) > 1000/cu.mm.
* No uncorrectable coagulopathy (INR>1.5, PTT and PT > 1.5 x the upper limit of normal)
* No uncorrectable thrombocytopenia (platelet count < 50,000/mm3)
* Life expectancy over 30 days
* RF ablation targets in the liver, lung or musculoskeletal system that meet the following criteria:

Hepatic lesions

* Intrahepatic metastases not amenable to other therapy
* Primary hepatic tumor if RF ablation of a portion of the tumor can lead to primary tumor resection rather than hepatic transplantation
* Single primary or multiple tumors in the liver
* At least one over 0.5 cm in diameter
* Edge of lesion not contiguous with main hepatic or common biliary duct.

Musculoskeletal lesions

* Local or regional recurrence of primary bone or soft tissue tumor not amenable to resection or radiotherapy
* Osseous, soft tissue or lymph node metastases not amenable to resection or radiotherapy.
* Head, neck, spine, extremity, chest wall, flank, abdominal wall, or pelvic bone or girdle lesions are treatable under this protocol
* RFA target < 50% of axial area in weight bearing bone unless reinforced with internal fixation (bone cement infusion) or in non-ambulatory patient.

Lung lesions

* No supplemental oxygenation is required.
* Metastatic solid tumor that has recurred or progressed after primary thoracotomy or thoracoscopic removal that is not amenable to radiotherapy, surgery or chemotherapy
* In the investigator's opinion, no supplemental oxygen will likely be required at rest for more than 30 days after RF ablation.
* Tumor burden < 20% of lung volume

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2003-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety of RFA in patients with childhood acquired tumors | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Krasin, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org